CLINICAL TRIAL: NCT07027995
Title: Food and Fitness With Medicine
Brief Title: Food and Fitness With Medicine (FFWM)
Acronym: FFWM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Colleen Spees, Professor of Medical Dietetics and Director of Hope Lab, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20250193
Record Dates: First submitted 2025-06-04; First posted 2025-06-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Kidney Metabolic Syndrome; Type 2 Diabetes
Keywords: Food is Medicine; Cardiovascular-kidney-metabolic; Exercise is Medicine; Post-menopausal Women; Medically Tailored Groceries; Type 2 Diabetes; Glucagon-like Peptide 1 Receptor Agonists; Nutrition; Behavior; GLP-1; Weight; Fitness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Behavior; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFWM+ (Experimental): Intervention Group receives medically tailored groceries and culinary training, fitness education and training, behavioral reinforcers, and access to a secure web portal.
  Interventions: Behavioral: Exercise is Medicine (EIM); Behavioral: Culinary Education; Behavioral: Food is Medicine; Behavioral: Nutrition Counseling; Behavioral: Participant Website
- Standard Care (No Intervention): Control Group - access to optional cooking demos

INTERVENTIONS:
Behavioral: Exercise is Medicine (EIM) — During Phase 1 (Weeks 1-12), participants are enrolled in a comprehensive 12-week fitness education and training program.
  Arms: FFWM+
Behavioral: Culinary Education — During Phase 1 & 2, participants receive monthly hybrid cooking demonstrations with culinary training.
  Arms: FFWM+
Behavioral: Food is Medicine — During Phase 1 (Weeks 1-12), participants receive bi-weekly medically tailored grocery vouchers.
  Arms: FFWM+
Behavioral: Nutrition Counseling — During Phase 1 (Weeks 1-12), participants engage in weekly behavioral nutrition counseling.
  Arms: FFWM+
Behavioral: Participant Website — During Phases 1 and 2, participants will receive digital behavioral reinforcers and access to a secure web portal that provides evidence-based resources.
  Arms: FFWM+

SUMMARY:
Food and Fitness with Medicine (FFWM) is a 24-week randomized controlled trial (RCT) enrolling 200 post-menopausal women (PMW) with stage 2 cardio-kidney metabolic (CKM) syndrome and type-2 diabetes (T2D) within 6 weeks of initiating glucagon-like peptide-1 receptor agonist (GLP-1RAs) to: 1. Examine discontinuation rates of GLP-1RAs (primary outcome); 2. Compare change in American Heart Association (AHA) PREVENT scores (secondary outcome); and 3. Examine the effects of FFWM on biologic mechanisms responsive to weight loss and cardiovascular health (CVH) including dermal carotenoids, body composition and metabolite biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of at least one of the following conditions: hypertension, type 2 diabetes, hyperlipidemia, chronic kidney disease, and/or metabolic syndrome.
* At least 18 years of age at the time of signing consent.
* Participants must have reliable transportation to attend Exercise is Medicine sessions.
* Access to an internet-enabled device.
* No objections to online grocery shopping, home food deliveries, or nutrition counseling.
* Residence meets Instacart delivery requirements (e.g., non-institutionalized).
* Participant is willing to use a personal credit card for Instacart back-up payments.
* Participants must speak English to be able to consent and engage in FIM and EIM programs.
* Participant has been clinically prescribed GLP-1RA's.

Exclusion Criteria:

* Conditions that impact digestion, metabolism, or food intake (e.g. surgical loss of esophagus, stomach, or colon, pancreatic dysfunction, bariatric surgery, brain surgery that alters cognition, etc.).
* Participants with uncontrolled mental illness disorders (e.g., schizophrenia, bipolar disorder, major depression, etc.) that are not well-managed or controlled through treatment, as determined by the study team.
* Familial history of certain cancers (e.g., multiple endocrine neoplasia, medullary thyroid carcinoma, etc.).
* Active digestive illnesses (i.e., Celiac disease, irritable bowel syndrome, chronic malabsorption).
* Comorbidities such as psychiatric or general illness that may put the subject at risk as determined by the investigator/s.
* Renal impairment, eGFR < 60 ml/min/1.73m2
* Factor which, in the investigator's opinion, is likely to compromise the subject's ability to participate in the study.
* Recent participation (e.g., 3 months) in other behavioral nutrition trials or programs (i.e., bariatric programs, diabetes education programs).
* Currently pregnant or planning to become pregnant during the study.
* Participant is not willing to provide a urine, blood, or stool sample.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants identified as post-menopausal females are eligible.
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
GLP-1 RA discontinuation rates | 0, 12, and 24 weeks
  GLP-1RA discontinuation rates will be captured using the electronic medical record to obtain medication name and formulation, dosage and frequency, prescription start and end dates, prescribing provider, refill information and prescription status (active, discontinued, completed), clinic notes or medication reconciliation fields confirming ongoing use or discontinuation, pharmacy records indicating medication pick-up (when available).

SECONDARY OUTCOMES:
American Heart Association (AHA) PREVENT Scores | 0, 12, and 24 weeks
  The AHA PREVENT scores are used in cardiovascular research to estimate the risk of future cardiovascular disease (CVD) based on factors such as BMI, age, sex, cholesterol, blood pressure, smoking, eGFR, diabetes, medication use, UACR, zip, and HbA1c. Scores are reported as a percent risk for CVD using the following scale: low (<5%), borderline (5% to 7.4%), itermediate (7.5% to 19.9%), and high (>20%).
Metabolites | 0, 12, and 24 weeks
  Stool and urine samples will be collected from participants to analyze metabolites at 3 study time points. Participants will collect samples and return within 7 days of a clinic visit. Samples will be processed and stored under strict biosafety protocols to maintain integrity.
Life's Essential 8 Scores | 0, 12, and 24 weeks
  The Life's Essential 8 Survey is a combination of questions used to assess and needed to accurately collect data to determine Life's essential 8 (LE8 scores for participants). Questions collect data on lifestyle health behaviors such as sleep patterns and smoking status. The Life's Essential 8 (LE8) is scored on a scale of 0 to 100. The LE8 score is used to assess and track an individual's overall cardiovascular health based on 8 key factors with a higher score indicating better cardiovascular health.
Blood Lipids | 0, 12, and 24 weeks
  Will be measured using Alere Cholestech LDX, respectively. We will perform a finger stick to obtain blood. The total amount of blood that will be collected for lipids (total cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL)) for this entire research study (3 time points over 24 weeks) is less than 2.5 mL (<1 teaspoon).
Body Composition | 0, 12, and 24 weeks
  We will look at body composition to monitor shifts in muscle mass, body fat, and visceral fat throughout the intervention. Participants will be weighed, wearing light clothing and without shoes, on a calibrated bioelectrical impedance scale (InBody 580) capable of analyzing body composition including visceral fat, total body fat percentage, lean body mass, and resting energy expenditure.
Dietary Patterns | 0, 12, and 24 weeks
  The National Cancer Institute's Dietary History Questionnaire (DHQIII) will be used to assess dietary patterns. The DHQIII tool is validated and assesses dietary intake of 134 foods and beverages in the past 30 days. Higher scores indicate better overall diet quality.
Hip Circumference | 0, 12, and 24 weeks
  Hip circumference will be measured with a measuring tape following the current NHANES Anthropometry Procedures Manual.
Dermal Carotenoid Scores | 0, 12, and 24 weeks
  Resonance Raman spectroscopy (RRS) is a non-invasive, validated method of measuring dermal carotenoids as a biomarker of fruit and vegetable intake. The Pharmanex NuSkin Biophotonic Scanner (model S3) uses a standardized RSS protocol intended for nutritional purposes and will not be used to diagnose any disease or medical condition. The scan involves passing a safe LED light across the surface of the skin for approximately 2 minutes. 2-3 measures will be obtained at each time point.
Blood Pressure | 0, 12, and 24 weeks
  Blood pressure including both systolic and diastolic blood pressure measures will be checked via an automated oscillometric sphygmomanometer (Omron 7 series).
Nutrition Security | 0, 12, 24 weeks.
  The Center for Nutrition and Health Impact Nutrition Security Screener will be used to assess nutrition security. The Center for Nutrition and Health Impact developed a four-item nutrition security screening tool. Three questions ask about household consumption and concerns around foods thought by the respondent to be good (or not) for health and well-being, and a fourth question asks about food variety.
Social and Emotional Wellbeing | 0, 12, and 24 weeks
  The De Jon Gierveld Social Isolation Scale will be used to asses social and emotional wellbeing. This short form, 6-item scale can be used as a reliable and valid measurement instrument for overall, emotional, and social loneliness. For this scale each item is assigned a score of 0 or 1 with the total possible score ranging form 0 to 6 with high scores indicating higher rates of loneliness.
Social Needs | 0, 12, and 24 weeks
  Centers for Medicare and Medicaid Services Accountable Health Communities Health-Related Social Needs Screening Tool will be used to identify needs. Tested by the CMS Innovation, this tool addresses the critical gap between clinical care and community services in the current health care delivery system by testing whether systematically identifying and addressing the health-related social needs of Medicare and Medicaid beneficiaries impacts their total health care costs and improves health. The questionnaire includes 26 questions addressing living situation, food security, transportation, utilities, safety, financial strain, employment, family and community support, education, physical activity, substance abuse, mental health and disabilities. This screening tool is not scored on a standardized scale rather participants screening positive for unmet social needs will be referred to available and free community resources (e.g., Health Impact Ohio, SNAP, MidOhio Food Farmacy, etc).
HbA1c | 0, 12, and 24 weeks
  Will be measured using Afinion 2 devices, respectively. We will perform a finger stick to obtain blood. The total amount of blood that will be collected for HbA1c for this entire research study (3 time points over 24 weeks) is less than 2.5 mL (<1 teaspoon).
Waist Circumference | 0, 12, and 24 weeks
  Waist circumference will be measured with a measuring tape following the current NHANES Anthropometry Procedures Manual.
Food Noise | 0, 12, 24 and weeks
  The Food Noise Questionnaire (FNQ) is a 5-item instrument to assess the frequency and intensity of intrusive food-related thoughts, urges, and preoccupations. Higher scores indicate greater perceived food noise.

OTHER OUTCOMES:
Household Size and Relationships | 0, 12, and 24 weeks
  PhenX Household Roster will be used to collect househol data. This survey requests participants to provide a list of all individuals currently residing in the household, starting with the person who owns or rents the dwelling (the householder), followed by the householder's spouse or partner, and then other household members. For each individual listed, the respondent will report their relationship to the householder and the householder's spouse, as well as their sex, age, and marital status.
Access to Healthcare | Baseline
  PhenX Health Insurance Coverage screener will be used to asses access to covergae. This brief survey includes questions designed to assess insurance coverage and health insurance type, in order to evaluate participant access to healthcare services.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen K Spees, PhD, MEd, RD, Principal Investigator — Ohio State University
Locations (4):
- United States (4):
  - Ohio State Healthy Community Center, Columbus, Ohio
  - Ohio State East Hospital, Columbus, Ohio
  - Martha Morehouse, Columbus, Ohio
  - Ohio State Outpatient Care Upper Arlington, Upper Arlington, Ohio

IPD SHARING:
Plan to Share IPD: No